CLINICAL TRIAL: NCT03602911
Title: A Comparison of NETSPOT Imaging Versus F-FDG-PET in Head and Neck Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1804059675
Record Dates: First submitted 2018-06-22; First posted 2018-07-27 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2023-06

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — gallium Ga 68 dotatate

STUDY DESIGN:
Intervention Model Description: Proof of Concept
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Proof of Concept (Other): The isotope 68Ga, available as NETSPOT and 18F-FDG-PET/CT per established protocol will both be administered
  Interventions: Drug: The isotope 68Ga, NETSPOT and 18F-FDG-PET/CT

INTERVENTIONS:
Drug: The isotope 68Ga, NETSPOT and 18F-FDG-PET/CT — All patients will undergo 18F-FDG-PET/CT per established protocol. Following 18F-FDG-PET/CT, the patient will undergo NETSPOT imaging

SUMMARY:
This is a proof-of-concept trial to compare 18F-FDG-PET/CT with NETSPOT (68Ga-DOTA-TATE), a commercially available radiotracer packet that utilizes 68Ga to image SSTR-specific tissue.

DETAILED DESCRIPTION:
Patients meeting inclusion criteria will be consented at the time of scheduling. All patients will undergo 18F-FDG-PET/CT per established protocol. Following 18F-FDG-PET/CT, the patient will undergo NETSPOT imaging with the AAA-provided dose. These scans will be performed no less than 8 hours, no more than 7 days apart. For patients undergoing same-day imaging, NETSPOT imaging will be performed prior to 18F-FDG-PET/CT. Following imaging, both 18F-FDG-PET/CT and NETSPOT imaging will be compared by trained neuroradiologists for SUV values and concordance with known sites of disease. Biopsies will be performed as is standard to verify all sites of primary or metastatic disease. Patients with oropharyngeal tumors will have HPV testing performed via the standard of care surrogate marker p16. Patients with p16-positive tumors will be recorded and analyzed separately for the above measures. Patients will be followed for a total of 1 year after the study and outcomes of overall survival, disease-free survival, presence and site of recurrence and development of metastatic disease will be recorded. All gathered data will be compared between reported 18F-FDG-PET/CT and NETSPOT imaging for true positive, true negative, positive predictive value and negative predictive value of patient groups.

ELIGIBILITY:
Inclusion Criteria:

Patients with suspected or diagnosed HNSCC undergoing planned 18F FDG PET/CT at the time of primary diagnosis or after completion of treatment.

Exclusion Criteria:

Inability to undergo 18F-FDG-PET/CT imaging due to medical comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rusha Patel, MD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University Medicine, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Proof of Concept
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Proof of Concept
Number analyzed (Participants) | 20
Age, Customized [Mean (Standard Deviation); unit: years] | 59.4 (11.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Detection and Staging of Head and Neck Squamous Cell Carcinoma Using Standard Uptake Value for NETSPOT Imaging
Description: NETSPOT imaging will be at least equivalent to 18F FDG PET/CT in the detection and staging of HNSCC. This will be done using Standard Uptake Value (SUV) measurements. SUV max of > 2.5 for 18F-FDG-PET and > 1.5 for 68GA DOTATATE-PET/CT were used as thresholds of concern.
  Using the PET scan, investigators calculated the standard uptake value (SUV), to compare the amount of an agent injected into the patient and the amount taken up by the tumor.
Time Frame: From Baseline up to day 7 post imaging
Measure: Median (Standard Deviation); unit: (SUV) volume (cm3)
Arm/Group | Proof of Concept
Number analyzed (Participants) | 20
(SUV) volume (cm3)
  OP-Primary Tumor | 7.21 (17.00)
  OP-Nodes | 4.84 (17.00)
  OC-Primary Tumor | 2.87 (17.00)
  OC-Nodes | 2.46 (17.00)
  Larynx-Nodes | 3.24 (17.00)

2. Secondary Outcome: Detection of Primary Site for Head and Neck Squamous Cell Carcinoma Using SUV Measurements With NETSPOT Imaging
Description: The Combination of NETSPOT imaging and 19F FDG PET/CT will have increased specificity for detecting the primary site for HNSCC of unknown primary than 18F FDG PET/CT alone. This will be done using Standard Uptake Value (SUV) measurements. SUV max of > 2.5 for 18F-FDG-PET and > 1.5 for 68GA DOTATATE-PET/CT were used as thresholds of concern.
  Using the PET scan, radiologists can calculate the standard uptake value (SUV), to compare the amount of an agent injected into the patient and the amount taken up by the tumor.
Time Frame: From Baseline up to day 7 post imaging
Measure: Median (Standard Deviation); unit: (SUV) volume (cm3)
Arm/Group | Proof of Concept
Number analyzed (Participants) | 20
(SUV) volume (cm3)
  OP-Primary Tumor | 14.98 (18.25)
  OP-Nodes | 7.59 (18.25)
  OC-Primary Tumor | 13.11 (18.25)
  OC-Nodes | 5.96 (18.25)
  Larynx-Nodes | 3.92 (18.25)

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Proof of Concept
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-12-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT03602911/Prot_SAP_003.pdf
  • Informed Consent Form (2017-12-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT03602911/ICF_004.pdf